CLINICAL TRIAL: NCT01449708
Title: Effect of Intraoperative Anesthetic Management on Postoperative Nausea and Vomiting (PONV) in Bariatric Surgery
Brief Title: Effect of Intraoperative Anesthetic Management on Postoperative Nausea and Vomiting in Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coastal Anesthesiology Consultants (Other)
Responsible Party: Principal Investigator, Patrick Ziemann-Gimmel, MD, Anesthesiologist, Principal Investigator, Coastal Anesthesiology Consultants
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3766 - 6886
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Bariatric Surgery; TIVA; PONV; non-opioid; OSA
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balanced Anesthesia (No Intervention): Patients will receive balanced general anesthesia including volatile anesthetics and narcotics. This reflects our current clinical practice.
- NoNarc TIVA (Active Comparator): Patients will receive narcotic free total intravenous anesthesia with Propofol, dexmedetomidine and ketamine
  Interventions: Drug: TIVA NoNarc

INTERVENTIONS:
Drug: TIVA NoNarc — * patients in both groups receive antiemetic prophylaxis
  * patients in the TIVA NoNarc group will receive propofol, dexmedetomidine, ketamine, ketorolac and acetaminophen intraoperatively
  * postop management in both groups is similar in both groups
  Arms: NoNarc TIVA

SUMMARY:
Morbidly obese patients are at high risk for Postoperative Nausea and Vomiting (PONV) after surgery and general anesthesia. The results of our observational study indicate that 42.7% of patients require medication to treat PONV in the first 24 hours after bariatric surgery despite our aggressive perioperative approach with triple prophylaxis. Common risk factors for PONV are the use of intraoperative narcotics and anesthetic gases.

Preliminary results of multimodal postoperative analgesia in the first 24 hours lead to a reduction of narcotic consumption, desaturations and use of antiemetic medication.

Our study hypothesis is that different types of anesthetics reduce PONV further.

Patient would be randomly assigned to receive either our current intraoperative management or a narcotic free, total intravenous general anesthetic (TIVA).

The investigators hope to improve patients' satisfaction by reducing PONV in the postoperative period.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for bariatric surgery at Flagler Hospital will be included after written and informed consent.

Exclusion Criteria:

* Patients will be excluded from the study if they don't consent to participate in the study. Patients allergic to any of the study medication will be excluded. Patients with second or third degree heart block will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ziemann-Gimmel, MD, Principal Investigator — Coastal Anesthesiology
Locations (1):
- Flagler Hospital, Saint Augustine, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziemann-Gimmel P, Goldfarb AA, Koppman J, Marema RT. Opioid-free total intravenous anaesthesia reduces postoperative nausea and vomiting in bariatric surgery beyond triple prophylaxis. Br J Anaesth. 2014 May;112(5):906-11. doi: 10.1093/bja/aet551. Epub 2014 Feb 18. PMID 24554545

RESULTS

PARTICIPANT FLOW:
Groups:
- Classic/Balanced Anesthesia: Patients will receive balanced general anesthesia including volatile anesthetics and narcotics. This reflects our current clinical practice. (Control)
  postop management in both groups is similar in both groups
- TIVA: TIVA NoNarc (Study): - patients in both groups receive antiemetic prophylaxis
  - patients in the TIVA NoNarc group will receive propofol, dexmedetomidine, ketamine, ketorolac and acetaminophen intraoperatively
Period: Overall Study
Arm/Group | Classic/Balanced Anesthesia | TIVA
Started | 61 | 63
Completed | 59 | 60
Not Completed | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — surgical complication | 1 | 2
Not completed — respiratory failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Classic/Balanced Anesthesia: Patients will receive balanced general anesthesia including volatile anesthetics and narcotics. This reflects our current clinical practice.
  * patients in both groups receive antiemetic prophylaxis
  * postop management in both groups is similar in both groups
- TIVA: * patients in both groups receive antiemetic prophylaxis
  * patients in the TIVA NoNarc group will receive propofol, dexmedetomidine, ketamine, ketorolac and acetaminophen intraoperatively
  * postop management in both groups is similar in both groups
- Total: Total of all reporting groups
Arm/Group | Classic/Balanced Anesthesia | TIVA | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (3.2) | 50.5 (3.5) | 50.4 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 16 | 21 | 37
Region of Enrollment [Number; unit: participants]
  United States | 59 | 60 | 119

OUTCOME MEASURES:

1. Primary Outcome: PONV During the First 24 Hours After Bariatric Surgery
Description: Postoperative Nausea and Vomiting
Time Frame: 24 hours
Measure: Number; unit: participants
Groups:
- Classic / Balanced Anesthesia: Patients will receive balanced general anesthesia including volatile anesthetics and narcotics. (Control)
- TIVA: patients in the TIVA NoNarc group will receive propofol, dexmedetomidine, ketamine, ketorolac and acetaminophen intraoperatively
Arm/Group | Classic / Balanced Anesthesia | TIVA
Number analyzed (Participants) | 59 | 60
participants | 22 | 12
Statistical Analysis 1: Comparison: Classic / Balanced Anesthesia vs TIVA; Test type: Superiority or Other; p = 0.04, Chi-squared; Relative Risk = 1.27, 95% CI 2-sided [1.01 to 1.61]

2. Secondary Outcome: Number of Patients Requiring Antiemetic Rescue Medication (AERM)
Time Frame: 24hours
Measure: Number; unit: participants
Arm/Group | Classic/Balanced Anesthesia | TIVA
Number analyzed (Participants) | 59 | 60
participants | 26 | 17

3. Secondary Outcome: PONV Between Different Surgical Procedures (Percentage of Participants)
Time Frame: 24 hours
Population: analysis was conducted with all participants and NOT per arm
Measure: Number; unit: percentage of participants
Groups:
- All Study Participants: measure included all119 patients depending on surgical procedure
Arm/Group | All Study Participants
Number analyzed (Participants) | 119
percentage of participants
  Sleeve Gastrectomy | 58.6
  Gastric Bypass (LRYGB) | 19.4
  Gastric Band | 0
  revision LRYGB | 23.1
  Conversion to LRYGB | 0
Statistical Analysis 1: Comparison: All Study Participants; Grouping of surgical procedures into three categories, analysis using bonferroni correction, 1) ReY group( gastric bypass, conversion to gastric bypass and revision gastric bypass) 2) Gastric Band (GB), 3) sleeve gastrectomy (SG); Test type: Superiority or Other; p = 0.009, Chi-squared; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.28 to 7.29]

ADVERSE EVENTS:
Time Frame: 24hours
Groups:
- Classic/Balanced Anesthesia: Patients will receive balanced general anesthesia including volatile anesthetics and narcotics. (Control)
Arm/Group | Classic/Balanced Anesthesia | TIVA
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No